CLINICAL TRIAL: NCT00052117
Title: A Phase 2, Randomized, Double-Blind, Dose-Ranging Study Of Capravirine (AG1549) In Combination With Kaletra (Trademark) and At Least 2 Nucleoside Reverse Transcriptase Inhibitors in Hiv-Infected Subjects Who Have Failed Antiretroviral Regimens Containing Protease Inhibitors, Nonnucleoside Reverse Transcriptase Inhibitors, and Nucleoside Reverse Transcriptase Inhibitors
Brief Title: Four-Drug Combination Treatment in Hiv-Infected Subjects Failing Therapy With Antiretroviral Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4311006
Record Dates: First submitted 2003-01-22; First posted 2003-01-23 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — capravirine; lopinavir-ritonavir drug combination

INTERVENTIONS:
Drug: capravirine
Drug: Kaletra
Drug: 2 NRTIs

SUMMARY:
This is a 48 week study for HIV-infected patients who have failed several regimens including PI's, NNRTs and NRTIs. Patients will be randomly selected to be in 1 of 4 groups. Three of the 4 groups will contain capravirine in different doses combined with Kaletra and nucleosides and one of the groups will be a combination of Kaletra and nucleosides without the capravirine.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected male or female at least 18 years of age
* HIV RNA level >1000 copies/mL at screening
* Subject has failed regimens that included at least 1 protease inhibitor but not more than 3 protease inhibitors, at least 1 nonnucleoside reverse transcriptase inhibitor, and least 2 nucleoside reverse transcriptase inhibitors
* Adequate renal function
* Adequate hematological function
* Adequate liver function

Exclusion Criteria:

* Women who are pregnant or lactating
* No previous experience with Kaletra

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-01; Study Completion 2005-05

PRIMARY OUTCOMES:
To determine the optimal safe and effective dose of capravirine in combination with Kaletra plus at least 2 NRTIs

SECONDARY OUTCOMES:
the relationship of HIV baseline resistance (genotype and phenotype) to virologic outcome
the population pharmacokinetics of capravirine and lopinavir/ritonavir (Kaletra) using mixed-effects modeling
the pharmacokinetic drug-drug interactions between capravirine and Kaletra and selected concomitant medications
changes in subject-reported health status and HIV symptoms using the Medical Outcomes Study - HIV Health Survey (MOS-HIV) and the Symptoms Distress Module (National Institute of Allergy and Infectious Diseases Adult AIDS Clinical Trials Group)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer